CLINICAL TRIAL: NCT03039166
Title: Metabolic and Structural Characterization of Hub's Vulnerability in Neurological Diseases Assessed by Ultra High Field Structural and Functional MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A01785-46; 2016-46 (Other: Assistance Publique-Hôpitaux de Marseille)
Record Dates: First submitted 2017-01-31; First posted 2017-02-01 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Diffuse Diseases
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- parkinson (Experimental)
  Interventions: Device: MRI 7T; Device: MRI 3 T
- partial epilepsy (Experimental)
  Interventions: Device: MRI 7T; Device: MRI 3 T
- alzheimer disease (Experimental)
  Interventions: Device: MRI 7T; Device: MRI 3 T
- multiple sclerosis (Experimental)
  Interventions: Device: MRI 7T; Device: MRI 3 T; Biological: blood sample
- amyotrophic lateral sclerosis (Experimental)
  Interventions: Device: MRI 7T; Device: MRI 3 T
- healthy control patients (Active Comparator)
  Interventions: Device: MRI 7T; Device: MRI 3 T

INTERVENTIONS:
Device: MRI 7T
Device: MRI 3 T
Biological: blood sample
  Arms: multiple sclerosis

SUMMARY:
the investigators hypothesize that hub alteration occurs both in diffuse diseases (MS, AD) as well as in more 'network specific' diseases (Parkinson, ALS, Epilepsy). This could impact on functional dysfunction not directly related to each disease, but that could induce common syndrome such as cognitive impairment observed in Parkinson, partial epilepsy or ALS.

The objective here is to test this hypothesis and provides better understandings on pathophysiological processes affecting those highly connected regions in 'diffuse' and 'focal' neurological diseases.

The ultimate goal is to identify new clinical targets for trans-nosological approaches (DBS, cognitive rehabilitation ...).

Practically, the investigators will explore 200 patients classified in 5 cohorts of 40 patients suffering for MS, AD, Parkinson, ALS, Epilepsy, using the last advanced methods to assess structural and functional brain connectivity implemented on the human 7T MR scanner equipping the CEMEREM (CHU Timone, Marseille, only 50 similar MR scanners worldwide).

In addition to high resolution diffusion MRI and rs-fMRI, metabolic and ionic (sodium) mapping will complement the MR protocol to characterize the pathophysiological processes of hub injury. Sixty healthy controls will also be explored wih the same protocol for normal database.

The proposal aims at characterizing and comparing from a morphological-functional point of view, the hub regions of patients suffering from these five diseases, to demonstrate the pertinence to preserve hub integrity as a major therapeutic target whatever the disease.

ELIGIBILITY:
Inclusion Criteria:

* Person female or male, more than 18-year-old,
* Person presenting unchecked general disease such as severe cancer, autoimmune disease, hepatic insufficiency, severe or untreated, shady arterial high blood pressure of the conduction or the disorder of the rhythm
* Person presenting chronic psychiatric disease, insane syndrome.
* Person presenting contraindication to the realization of an examination by MRI (metallic claustrophobia, foreign body, pacemakers),
* Person benefiting from a social security cover,
* Person having read, understood and signed an informed consent after information

Exclusion Criteria:

* Claustrophobia,
* Metallic foreign bodies,
* Pacemakers,
* Severe renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2022-02 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Index of reorganization of the structural hubs (ks-Degree) | 5years

SECONDARY OUTCOMES:
Concentrations of sodium within hubs | 5 years
Concentrations of Glutamate/Glutamine within hubs | 5 years
cortical Thicknesses within hubs | 5 years
Iron accumulation within hubs | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Catherine GEINDRE, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assiatnce Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No